CLINICAL TRIAL: NCT06726772
Title: Post-COVID-19 Symptom Burden: Effects of an Outpatient Group Psychotherapy in Long COVID Patients
Brief Title: Group Psychotherapy in Long COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Katja Haemmerli Keller, Head Psychologist, Cantonal Hospital of St. Gallen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSOMA-2022-4
Record Dates: First submitted 2024-12-06; First posted 2024-12-10 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Long COVID; COVID-19
Keywords: COVID-19; Long COVID; Long COVID-19 Syndrome; Group Psychotherapy; Cognitive Behavioral Therapy; CBT; Acceptance and Commitment Therapy; ACT; Psychometrics
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19 | interventions — Psychotherapy, Group

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Group Psychotherapy) (Experimental)
  Interventions: Behavioral: Group Psychotherapy

INTERVENTIONS:
Behavioral: Group Psychotherapy — Group psychotherapy based on Cognitive Behavioral Therapy (CBT) and Acceptance and Commitment Therapy (ACT) elements

SUMMARY:
The aim of the present study was to establish a single-arm group psychotherapy and to evaluate its clinical effectiveness in long COVID patients.

DETAILED DESCRIPTION:
This study took place at the Cantonal Hospital St.Gallen, a tertiary care hospital in Eastern Switzerland, and included data collection between November 2021 and January 2024. During this time span, the same licensed psychotherapist conducted the group psychotherapy six times in total with a maximum of nine patients each. Each of the six groups had one-hour group therapy sessions weekly within eight consecutive weeks. During the study period, the group psychotherapy was part of a more comprehensive treatment for long COVID as all patients primarily received active pacing therapy.

The investigators implemented cognitive-behavioral therapy (CBT) and acceptance and commitment therapy (ACT) elements into group psychotherapy and focused on fatigue, insomnia, depression, anxiety, somatic symptoms, psychotraumatology, and quality of life as psychosomatic outcome measures (pre- and post-interventional).

ELIGIBILITY:
Inclusion Criteria:

* Signed general consent form of the Cantonal Hospital of St.Gallen
* Adult patients (≥ 18 years of age)
* Long COVID diagnosis made as part of the long COVID consultation at the Cantonal Hospital of St.Gallen
* Screening for psychological stress and suitability for group therapy through an initial consultation with a psychotherapeutic specialist from the Department of Psychosomatic Medicine and Consultation-Liaison Psychiatry at the Cantonal Hospital of St.Gallen

Exclusion Criteria:

* Insufficient language skills for completing the questionnaires in German
* Refusal to sign the general consent form
* Severe mental disorders requiring an individualized setting, i.e. suicidal tendencies at the time of screening, acute psychosis and personality disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Change of Fatigue Score measured with the Questionnaire "FSS" (Fatigue Severity Scale) from baseline to 8 weeks | From enrollment to the end of treatment at 8 weeks
  9 is equivalent to no fatigue and 63 indicates the worst possible fatigue.
Change of Insomnia Score measured with the Questionnaire "ISI" (Insomnia Severity Index) from baseline to 8 weeks | From enrollment to the end of treatment at 8 weeks
  0 is equivalent to no insomnia and 28 indicates the worst possible insomnia.
Change of Quality of Life and Current Health Status measured with the Questionnaire "EQ-5D-5L" (European Quality of Life 5 Dimensions 5 Level Version) from baseline to 8 weeks | From enrollment to the end of treatment at 8 weeks
  0 (and -0.59) is equivalent to the lowest quality of life (and current health) and 100 (and 1) indicates the best possible quality of life (and current health)
Change of Depression and Anxiety Score measured with the Questionnaire "HADS" (Hospital Anxiety and Depression Scale) from baseline to 8 weeks | From enrollment to the end of treatment at 8 weeks
  0 is equivalent to no depression/anxiety and 21 indicates the worst possible depression/anxiety.
Change of Depression, Anxiety, and Somatic Symptom Scores measured with the Questionnaire "PHQ-SADS" (Patient Health Questionnaire) from baseline to 8 weeks | From enrollment to the end of treatment at 8 weeks
  0 is equivalent to no depression/anxiety/somatic symptoms and 30 indicates the worst possible depression/anxiety/somatic symptoms.
Change of Psychotraumatology Score measured with the Questionnaire "IES-R" (Impact of Event Scale-revised) from baseline to 8 weeks | From enrollment to the end of treatment at 8 weeks
  -4.36 is equivalent to no psychotraumatology (no suspected PTSD) and 2.99 indicates the worst possible psychotraumatology (suspected PTSD). A score equally or greater than zero (cut-off point) indicates suspected PTSD.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychosomatic Medicine and Consultation-Liaison Psychiatry, Cantonal Hospital St.Gallen, Switzerland, Sankt Gallen, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available from the corresponding author upon reasonable request.